CLINICAL TRIAL: NCT01549054
Title: A Single-center, Randomized, Open-label, Two-part Study to Evaluate Bioavailability of Prototype Third-generation Formulations of E5501 Relative to Second-generation Tablet Formulation in Healthy Subjects
Brief Title: A Study in Healthy Subjects to Evaluate Bioavailability of 4 Formulations of E5501
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E5501-G000-012
Record Dates: First submitted 2012-01-31; First posted 2012-03-08 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10-mg dose of E5501 2G tablet (Experimental)
  Interventions: Drug: 10-mg dose of E5501 2G tablet
- 10-mg dose of E5501 cyclodextrin oral solution (Experimental)
  Interventions: Drug: 10-mg dose of E5501 cyclodextrin oral solution
- 10-mg dose of E5501-P21% powder (Experimental)
  Interventions: Drug: 10-mg dose of E5501-P21% powder
- 10-mg dose of E5501 lipid-based oral (Experimental)
  Interventions: Drug: 10-mg dose of E5501 lipid-based oral

INTERVENTIONS:
Drug: 10-mg dose of E5501 2G tablet — Treatment A: Single 10-mg dose of E5501 2G tablet
  Arms: 10-mg dose of E5501 2G tablet
Drug: 10-mg dose of E5501 cyclodextrin oral solution — Treatment B: Single 10-mg dose of E5501 cyclodextrin oral solution
  Arms: 10-mg dose of E5501 cyclodextrin oral solution
Drug: 10-mg dose of E5501-P21% powder — Treatment C: Single 10-mg dose of E5501-P21% powder oral suspension
  Arms: 10-mg dose of E5501-P21% powder
Drug: 10-mg dose of E5501 lipid-based oral — Treatment D: Single 10-mg dose of E5501 lipid-based oral suspension
  Arms: 10-mg dose of E5501 lipid-based oral

SUMMARY:
This is a study in healthy subjects. There are two parts to the study. In the first part of the study each subject will receive a single 10mg dose of each of the four formulations of E550. Based on the results from Part 1, an optimal formulation will be selected for further evaluation in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women (age ≥ 18 to ≤ 55 years)
* Body mass index ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2 at the time of screening and baseline of Treatment Period 1
* Platelet count between 120 x 109/L and 300 x 109/L at baseline of each Treatment Period 1, 3, and 5
* Women of child bearing potential must agree to use a highly effective method of contraception, other than estrogen-based hormonal contraceptives, during the Treatment Phase of the study.

In addition, other standard criteria for healthy subjects will be used.

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact the PK of study drug
* Agents associated with thrombotic events (including oral contraceptives) must be discontinued within 30 days of first study drug administration
* Evidence of organ dysfunction or any clinically significant event or illness in the subject's medical history, e.g., history of splenectomy.
* History of arterial or venous thrombosis, including partial or complete thrombosis (e.g., stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism). Known family history of hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency, etc.)
* Hemoglobin less than the lower limit of normal levels.

In addition, other standard criteria for healthy subjects will be used.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentrations of drug for each dose over time as measured by AUC, CMAX, TMax | 133 days

SECONDARY OUTCOMES:
Change in plasma concentrations of drug for each dose over time as measured by AUC, CMAX, TMax with and without food | 133 days

CONTACTS AND LOCATIONS:
Overall Officials: Bhaskar Rege, Study Director — Eisai Inc.
Locations (1):
- Quotient, Nottingham, United Kingdom